CLINICAL TRIAL: NCT01517191
Title: Sentinel Surveillance for Influenza Requiring Hospital Admission Canadian Adults
Acronym: SOS-VE01
Status: Completed | Type: Observational
Sponsor: Dalhousie University (Other)
Collaborators: Public Health Agency of Canada (PHAC) (Other Government); Canadian Institutes of Health Research (CIHR) (Other Government); GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: SOS-VE01
Record Dates: First submitted 2012-01-17; First posted 2012-01-25 (Estimated); Last update posted 2018-03-30 (Actual); Status verified 2018-03

CONDITIONS: Influenza
Keywords: Influenza; Respiratory Infection
MeSH Terms: conditions — Influenza, Human; Respiratory Tract Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum and Nasopharyngeal swabs
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Influenza Positive Case: Influenza cases are hospitalized adults who have tested positive for influenza.
- Influenza Negative Control: Control Controls are hospitalized adults who have tested negative for influenza.

SUMMARY:
This surveillance study will include all consenting adults hospitalized with influenza (cases) at the SOS network of hospitals as well as influenza negative patients(controls), to assess vaccine effectiveness in each group. Both groups will be followed throughout their hospitalization and for 30 days post discharge to monitor severity of illness and outcomes following their illness.

DETAILED DESCRIPTION:
The Canadian Immunization Research Network(CIRN) is a collaborative research network which brings together over 100 investigators in over 40 institutions to evaluate all factors relevant to the introduction of a pandemic influenza vaccine in Canada. The Serious Outcomes Surveillance (SOS) Network within CIRN was established in 2009 to plan for evaluation of influenza vaccine safety and effectiveness. Vaccine effectiveness studies are critical in assessing vaccine effectiveness under real world conditions and in assessing vaccine effectiveness in the prevention of severe outcomes. Establishing the methodology and infrastructure for real-time field assessment of vaccine effectiveness is crucial to inform policy recommendations for the optimal use of resources, including vaccines.

This study will include all consenting adult patients hospitalized at one of the SOS Network hospitals during influenza season who test positive for influenza (cases). In addition two influenza negative controls will be matched to each case to measure differences in vaccine effectiveness. Specific study aims are:

1. To determine the effectiveness of trivalent influenza vaccination (TIV in general, and GSK TIV in particular) in preventing influenza-associated hospitalization in adults ≥ 65 years,
2. To determine the effectiveness of influenza vaccination in preventing influenza-associated death in adults ≥ 65 years
3. To determine the effectiveness of influenza vaccination in preventing influenza-associated hospitalization and death in adults < 65 years
4. To characterize the burden of disease, clinical outcomes, and resource utilization associated with influenza A and influenza B lineages
5. To examine clinical and immunologic factors impacting on severity of disease and influenza vaccine effectiveness in adults

ELIGIBILITY:
Inclusion Criteria:

* Adult patients ≥ 16 years of age admitted to participating SOS Network hospitals with the following admitting diagnoses will be eligible for screening:
* pneumonia
* acute exacerbation of chronic obstructive pulmonary disease (AECOPD) or asthma
* unexplained sepsis
* Any other respiratory infection or diagnosis Or any respiratory or influenza-like symptom )(eg dyspnea, cough, sore throat, myalgia, arthralgia, fever, delirium/altered level of consciousness, CHF)

Exclusion Criteria:

* Patients whose reason for admission was clearly unrelated to the presence of influenza (for example, patients admitted due to trauma, elective surgery, or patients who have an alternative diagnosis that is clearly not respiratory,, e.g. cellulitis, intra-abdominal process, or gastrointestinal bleeding) Unless being enrolled as a nosocomial influenza case
* Patients whose onset of symptoms was prior to or within 72 hours of hospital admission but who were not tested for influenza within 7 days of hospital admission. These should be captured on the screening form as screen failures.
* No children in care will be enrolled in the study

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This observational study is open to adults admitted to hospital with test postitive influenza or with an influenza like illness who test negative.
Sampling Method: Probability Sample
Enrollment: 4197 (Actual)
Dates: Start 2011-11; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Estimate the burden of influenza disease and influenza vaccine effectiveness. | 1 Year
  Occurrence of any PCR-confirmed influenza virus infection in vaccinated (>14 days after receipt of seasonal influenza vaccine) or unvaccinated adults ≥ 65 years of age.

SECONDARY OUTCOMES:
Estimate the burden of influenza disease and influenza vaccine effectiveness. | 1 Year
  Occurrence of any PCR-confirmed influenza virus infection in vaccinated (>14 days after receipt of seasonal influenza vaccine) or unvaccinated adults ≥ 16 years of age

CONTACTS AND LOCATIONS:
Overall Officials: Shelly A McNeil, MD, Principal Investigator — Dalhousie University
Locations (14):
- Canada (14):
  - Vancouver General, Vancouver, British Columbia
  - The Moncton Hospital, Moncton, New Brunswick
  - Saint John Regional Hospital, Saint John, New Brunswick
  - QEII Health Science Centre, Halifax, Nova Scotia
  - William Osler Health Center, Brampton, Ontario
  - Advanced Medical Research Institue of Canada, Greater Sudbury, Ontario
  - McMaster, Hamilton, Ontario
  - Ottawa General, Ottawa, Ontario
  - North York General Hospital, Toronto, Ontario
  - Toronto East General Hospital, Toronto, Ontario
  - Mount Sinai, Toronto, Ontario
  - MUCH, Montreal, Quebec
  - CHUS, Sherbrooke, Quebec
  - CHUl/CHUQ, Québec

REFERENCES:
- [Derived] Pott H, LeBlanc JJ, ElSherif M, Hatchette TF, Andrew MK, McNeil SA. Human Metapneumovirus Epidemiology Among Middle-aged and Older Adults Hospitalized With Acute Respiratory Infection. J Infect Dis. 2025 Jul 16;232(Supplement_1):S69-S77. doi: 10.1093/infdis/jiaf083. PMID 40668096
- [Derived] Pott H, Andrew MK, Shaffelburg Z, Nichols MK, Ye L, ElSherif M, Hatchette TF, LeBlanc JJ, Ambrose A, Boivin G, Bowie W, Johnstone J, Katz K, Lagace-Wiens P, Loeb M, McCarthy A, McGeer A, Poirier A, Powis J, Richardson D, Semret M, Smith S, Smyth D, Stiver G, Trottier S, Valiquette L, Webster D, McNeil SA. Oseltamivir Reduces 30-Day Mortality in Older Adults With Influenza: A Pooled Analysis From the 2012-2019 Serious Outcomes Surveillance Network of the Canadian Immunization Research Network. Open Forum Infect Dis. 2025 Feb 3;12(2):ofaf058. doi: 10.1093/ofid/ofaf058. eCollection 2025 Feb. PMID 39968306
- [Derived] Shoukat A, Bawden CE, Rost G, LeBlanc JJ, Galvani AP, Langley JM, Moghadas SM. Impact and cost-effectiveness analyses of vaccination for prevention of respiratory syncytial virus disease among older adults in Ontario: A Canadian Immunization Research Network (CIRN) study. Vaccine. 2024 Mar 7;42(7):1768-1776. doi: 10.1016/j.vaccine.2024.02.041. Epub 2024 Feb 16. PMID 38368226
- [Derived] Mulpuru S, Andrew MK, Ye L, Hatchette T, LeBlanc J, El-Sherif M, MacKinnon-Cameron D, Aaron SD, Alvarez GG, Forster AJ, Ambrose A, McNeil SA; Serious Outcomes Surveillance and Canadian Immunization Research Network (CIRN) Investigators. Impact of respiratory viral infections on mortality and critical illness among hospitalized patients with chronic obstructive pulmonary disease. Influenza Other Respir Viruses. 2022 Nov;16(6):1172-1182. doi: 10.1111/irv.13050. Epub 2022 Sep 7. PMID 36069141
- [Derived] LeBlanc JJ, ElSherif M, Mulpuru S, Warhuus M, Ambrose A, Andrew M, Boivin G, Bowie W, Chit A, Dos Santos G, Green K, Halperin SA, Hatchette TF, Ibarguchi B, Johnstone J, Katz K, Langley JM, Lagace-Wiens P, Loeb M, Lund A, MacKinnon-Cameron D, McCarthy A, McElhaney JE, McGeer A, Poirier A, Powis J, Richardson D, Semret M, Shinde V, Smyth D, Trottier S, Valiquette L, Webster D, Ye L, McNeil SA. Validation of the Seegene RV15 multiplex PCR for the detection of influenza A subtypes and influenza B lineages during national influenza surveillance in hospitalized adults. J Med Microbiol. 2020 Feb;69(2):256-264. doi: 10.1099/jmm.0.001032. Epub 2019 Jun 28. PMID 31264957
- [Derived] Mulpuru S, Li L, Ye L, Hatchette T, Andrew MK, Ambrose A, Boivin G, Bowie W, Chit A, Dos Santos G, ElSherif M, Green K, Haguinet F, Halperin SA, Ibarguchi B, Johnstone J, Katz K, Langley JM, LeBlanc J, Loeb M, MacKinnon-Cameron D, McCarthy A, McElhaney JE, McGeer A, Powis J, Richardson D, Semret M, Shinde V, Smyth D, Trottier S, Valiquette L, Webster D, McNeil SA; Serious Outcomes Surveillance (SOS) Network of the Canadian Immunization Research Network (CIRN). Effectiveness of Influenza Vaccination on Hospitalizations and Risk Factors for Severe Outcomes in Hospitalized Patients With COPD. Chest. 2019 Jan;155(1):69-78. doi: 10.1016/j.chest.2018.10.044. PMID 30616737
- [Derived] Nichols MK, Andrew MK, Ye L, Hatchette TF, Ambrose A, Boivin G, Bowie W, Dos Santos G, Elsherif M, Green K, Haguinet F, Katz K, Leblanc J, Loeb M, MacKinnon-Cameron D, McCarthy A, McElhaney JE, McGeer A, Powis J, Richardson D, Semret M, Sharma R, Shinde V, Smyth D, Trottier S, Valiquette L, Webster D, McNeil SA; Serious Outcomes Surveillance (SOS) Network of the Canadian Immunization Research Network (CIRN). The Impact of Prior Season Vaccination on Subsequent Influenza Vaccine Effectiveness to Prevent Influenza-related Hospitalizations Over 4 Influenza Seasons in Canada. Clin Infect Dis. 2019 Aug 30;69(6):970-979. doi: 10.1093/cid/ciy1009. PMID 30508064
- [Derived] Nichols MK, Andrew MK, Hatchette TF, Ambrose A, Boivin G, Bowie W, Chit A, Dos Santos G, ElSherif M, Green K, Haguinet F, Halperin SA, Ibarguchi B, Johnstone J, Katz K, Lagace-Wiens P, Langley JM, LeBlanc J, Loeb M, MacKinnon-Cameron D, McCarthy A, McElhaney JE, McGeer A, Poirier A, Powis J, Richardson D, Schuind A, Semret M, Shinde V, Smith S, Smyth D, Stiver G, Taylor G, Trottier S, Valiquette L, Webster D, Ye L, McNeil SA; Serious Outcomes Surveillance Network of the Canadian Immunization Research Network (CIRN), the Toronto Invasive Bacterial Diseases Network (TIBDN). Influenza vaccine effectiveness to prevent influenza-related hospitalizations and serious outcomes in Canadian adults over the 2011/12 through 2013/14 influenza seasons: A pooled analysis from the Canadian Immunization Research Network (CIRN) Serious Outcomes Surveillance (SOS Network). Vaccine. 2018 Apr 12;36(16):2166-2175. doi: 10.1016/j.vaccine.2018.02.093. Epub 2018 Mar 13. PMID 29548608
- [Derived] Andrew MK, Shinde V, Hatchette T, Ambrose A, Boivin G, Bowie W, Chit A, Dos Santos G, ElSherif M, Green K, Haguinet F, Halperin SA, Ibarguchi B, Johnstone J, Katz K, Langley JM, LeBlanc J, Loeb M, MacKinnon-Cameron D, McCarthy A, McElhaney J, McGeer A, Nichols MK, Powis J, Richardson D, Semret M, Stiver G, Trottier S, Valiquette L, Webster D, Ye L, McNeil SA; Public Health Agency of Canada/Canadian Institutes of Health Research Influenza Research Network (PCIRN) Serious Outcomes Surveillance Network and the Toronto Invasive Bacterial Diseases Network (TIBDN). Influenza vaccine effectiveness against influenza-related hospitalization during a season with mixed outbreaks of four influenza viruses: a test-negative case-control study in adults in Canada. BMC Infect Dis. 2017 Dec 29;17(1):805. doi: 10.1186/s12879-017-2905-8. PMID 29284435
- [Derived] Andrew MK, Shinde V, Ye L, Hatchette T, Haguinet F, Dos Santos G, McElhaney JE, Ambrose A, Boivin G, Bowie W, Chit A, ElSherif M, Green K, Halperin S, Ibarguchi B, Johnstone J, Katz K, Langley J, Leblanc J, Loeb M, MacKinnon-Cameron D, McCarthy A, McGeer A, Powis J, Richardson D, Semret M, Stiver G, Trottier S, Valiquette L, Webster D, McNeil SA; Serious Outcomes Surveillance Network of the Public Health Agency of Canada/Canadian Institutes of Health Research Influenza Research Network (PCIRN) and the Toronto Invasive Bacterial Diseases Network (TIBDN). The Importance of Frailty in the Assessment of Influenza Vaccine Effectiveness Against Influenza-Related Hospitalization in Elderly People. J Infect Dis. 2017 Aug 15;216(4):405-414. doi: 10.1093/infdis/jix282. PMID 28931244